CLINICAL TRIAL: NCT03669848
Title: Is Transcutaneous Carbon Monoxide Saturation of E-cigarette Users Comparable to That of Smokers?
Acronym: COVAP
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI18 / COVAP; 2018-A01471-54 (Other: IdRCB)
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Carbon Monoxide Poisoning
Keywords: carbon monoxide poisoning; e-cigarette user; transcutaneous saturation measurements
MeSH Terms: conditions — Carbon Monoxide Poisoning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulse CO-oximetry: Measuring blood Carbon Monoxide levels with Pulse CO-oximetry (SpCO) Measurements are taken with a noninvasive method by placing a sensor on a patient, usually on the fingertip.
  Interventions: Other: Pulse CO-oximetry

INTERVENTIONS:
Other: Pulse CO-oximetry — Measuring blood Carbon Monoxide levels with Pulse CO-oximetry (SpCO)

SUMMARY:
Suspicions of carbon monoxide poisoning that lead to the treatment of victims are numerous. Measurement of transcutaneous carbon monoxide saturation (SpCO) is a useful diagnostic and triage tool for victims and the toxic threshold is clearly defined for both non-smokers (SpCO> 5%) and smokers ( SpCO> 10%).

Currently, the use of e-cigarettes is democratizing. Unfortunately, the threshold for toxic SpCO is not defined for this patient profile.

The risk is treating in excess or worse than underestimating carbon monoxide poisoning in e-cigarette users who would be exposed to carbon monoxide exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to adult emergency department
* Age ≥ 18 years

Exclusion Criteria:

* Passive exposure to tobacco
* Mixed exposure (tobacco / e-cigarette)
* Patient having objected to the processing of his data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active smoker presenting to adult emergency department
Sampling Method: Non-Probability Sample
Enrollment: 1116 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Blood Carbon Monoxide levels measurements | Baseline
  Measuring blood Carbon Monoxide levels with Pulse CO-oximetry (SpCO)

CONTACTS AND LOCATIONS:
Overall Officials: Leila CAMBONI, MD, Principal Investigator — University Hospital, Tours
Locations (1):
- Adult Emergency Department, University Hospital, Tours, Tours, France